CLINICAL TRIAL: NCT03578731
Title: Efficacy of the "Consilium" Smartphone App for Detecting Symptoms and Treatment Side Effects in Cancer Patients Depending on Form of Medication Application, Age and Outpatient Characteristics: Observational Study
Brief Title: Efficacy of the "Consilium" Smartphone App for Detecting Symptoms and Treatment Side Effects in Cancer Patients
Acronym: APP-2
Status: Terminated | Type: Observational
Why Stopped: Mainly due to insufficient recruitment
Sponsor: OnkoZentrum Zürich AG (Other)
Collaborators: Stiftung Swiss Tumor Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-02028
Record Dates: First submitted 2018-05-08; First posted 2018-07-06 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2020-11

CONDITIONS: Telemedicine; eHealth
Keywords: APP; ePRO; electronic patient reported outcome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Consilium-APP: Patients with oncological, medical treatment for breast cancer, colon cancer, prostate cancer, lung cancer or hematological malignancies.
  Interventions: Device: app

INTERVENTIONS:
Device: app — The app is used to record the study parameters for a period of 90 days.
  The following measures are used for data collection:
  * Interview during regular consultation with doctor
  * Web-App for gathering doctors data
  * "Consilium" Smartphone App for gathering patient data During the course of care, the patient enters in a regular manner symptoms and treatment side effects in the Smartphone app. A continuous capture of the symptoms and treatment side effect is provided. If no entry is made within 3 days the patient is prompted to enter the data via a push message.
  * Well-being through a patient rating on a visual analog scale
  * Registration of symptoms and treatment side effects is done through the app
  After completion of the study patients will be questioned according to:
  • Usability and usefulness of the Smartphone app

SUMMARY:
The study investigates the influence of the use of a Smartphone App, on changes in general well-being and the occurrence of symptoms during a tumor therapy. With this documentation, medical professionals should be enabled to judge the influence of symptoms on quality of life during different time periods, between planed visits on site.

DETAILED DESCRIPTION:
The study will examine the number, characteristics and intensity of electronically reported symptoms and therapy side effects depending on treatment and characteristics of patients with cancer of breast, colon, prostate, lung and hematological malignancies during a three-month period from the initiation of therapy. This period frequently represents the duration of a therapeutic regimen.

The level of agreement κ between the ECOG/CTCAE ratings by physicians at the time of the regular consultation, and the ratings derived from the daily PROs between consultations, will be analyzed in order to determine the reliability and utility of self-reported electronic symptom monitoring.

The purpose is to evaluate different qualities of symptoms self-reported electronically between consultations with respect to the course of treatment application, out-patient settings, gender and age. In particular, outpatients with frequent (weekly) consultations will be compared to patients with infrequent consultations (3-weekly or less frequent).

The study will also aim to identify the conditions and factors that might increase the likelihood of an unplanned consultation or emergency hospitalization.

In particular, the proposed study design and associated primary and secondary endpoints will enable us to test the following hypotheses:

1. In patient groups with infrequent outpatient visits (3-weekly or less) as is determined by the treatment schedule, the level of agreement κ between ePRO-derived ECOG/CTCAE ratings and physician-derived ECOG/CTCAE ratings (at time of consultation) is at least as high as in patient groups with weekly visits for symptoms having occurred within the week before the visit. However, κ is expected lower in the group with infrequent visits for symptoms having occurred more than 2 weeks prior to consultation, due to higher fidelity of ePRO-derived ratings for long-ago symptoms.
2. Regular visits of outpatients undergoing infusion therapy (as determined by the treatment schedule) do not significantly decrease the number of unplanned and emergency consultations necessary.
3. Young female and older male patient groups report significantly more severe and worsening symptoms and side effects.

Patients with the most common types of cancer in the treatment center will be included:

Breast, Colon, Prostate, Lung, Hematological malignancies

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Women or men aged ≥ 18 years
* Patients with breast, colon, prostate, lung cancer or hemat. malignancies
* Initiation or change of therapy for the types of cancer mentioned above
* German speaking
* Personal smartphone with iOS or Android system

Exclusion Criteria:

* Patients whose compliance must be questioned, e.g. due to a psychological disorders or private life situation
* Patients with insufficient knowledge of smartphone use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with the most common types of cancer in the treatment center will be included: Breast, Colon, Prostate, Lung, Hematological malignancies
Sampling Method: Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2020-10-10 (Actual); Study Completion 2020-10-10 (Actual)

PRIMARY OUTCOMES:
Level of agreement | 12 weeks of treatment
  Level of agreement κ with respect to categories of common toxicity criteria (ECOG/CTCAE) categories between ePRO recording and the treating physician at time of consultation

SECONDARY OUTCOMES:
ePRO and therapy side effects | 12 weeks of treatment
  Assessment of the number, characteristics and intensity of electronically reported symptoms and therapy side effects during the first three months of therapy
Rating of different qualities of electronically reported symptoms in out-patient settings | 12 weeks of treatment
  Rating of different qualities of electronically reported symptoms in out-patient settings with respect to: course of treatment application (oral vs. infusion vs. radiation), treatment (systemic vs. local), gender and age
Unplanned consultations | 12 weeks of treatment
  Number and nature of unplanned consultations, (consultation vs. emergency hospitalizations)
Hospital days | 12 weeks of treatment
  Number of days in the hospital during for each event (≤2 days or > 2 days)
Patient characteristics for discontinued use of mobile monitoring | 12 weeks of treatment
  Assessment of patients' characteristics for a discontinuation of the use of the mobile monitoring
Usability and usefulness of smartphone app | 12 weeks of treatment
  Evaluation of the usability and usefulness of the smartphone app in the course of the treatment as rated by physician and patient after completion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Trojan, Prof. Dr. med., Principal Investigator — OnkoZentrum Zürich AG
Locations (18):
- LKH Feldkirch, Innere Medizin II, Feldkirch, Austria
- Germany (3):
  - Universitätsklinikum Halle (Saale) Universitätsklinik und Poliklinik für Gynäkologie, Halle
  - Universitätsklinikum Schleswig-Holstein, Klinik für Frauenheilkunde und Geburtshilfe (Gynäkologie), Lübeck
  - Sana Klinikum Offenbach Abteilung Gynäkologie und Geburtshilfe, Offenbach
- Switzerland (14):
  - OnkoZentrum Zürich AG, Zurich, Canton of Zurich
  - Kantonsspital Aarau, Aarau
  - Tumor Zentrum Aarau - Hirslanden Medical Center, Aarau
  - Onkologie Praxis Lindenhofspital, Bern
  - PROLINDO - Lindenhofspital, Bern
  - Oncocare Klinik Engeried, Bern
  - TUCARE, Bülach
  - Onko-Hämatologisches Zentrum Zug, Cham
  - Kantonsspital Baselland, Liestal
  - Limmattal Spital, Schlieren
  - Onkologiepraxis Bellvue, Zurich
  - Brust-Zentrum Zürich, Zurich
  - OnkoZentrum Hirslanden, Zurich
  - Universitätsspital Zürich, Klinik für Gynäkologie, Zurich

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: 2020/2021
URL: https://www.clinicaltrials.gov/ct2/search

REFERENCES:
- [Derived] Trojan A, Kuhne C, Kiessling M, Schumacher J, Drose S, Singer C, Jackisch C, Thomssen C, Kullak-Ublick GA. Impact of Electronic Patient-Reported Outcomes on Unplanned Consultations and Hospitalizations in Patients With Cancer Undergoing Systemic Therapy: Results of a Patient-Reported Outcome Study Compared With Matched Retrospective Data. JMIR Form Res. 2024 May 6;8:e55917. doi: 10.2196/55917. PMID 38710048
- [Derived] Trojan A, Roth S, Atassi Z, Kiessling M, Zenhaeusern R, Kadvany Y, Schumacher J, Kullak-Ublick GA, Aapro M, Eniu A. Comparison of the Real-World Reporting of Symptoms and Well-Being for the HER2-Directed Trastuzumab Biosimilar Ogivri With Registry Data for Herceptin in the Treatment of Breast Cancer: Prospective Observational Study (OGIPRO) of Electronic Patient-Reported Outcomes. JMIR Cancer. 2024 Apr 4;10:e54178. doi: 10.2196/54178. PMID 38573759
- [Derived] Trojan A, Leuthold N, Thomssen C, Rody A, Winder T, Jakob A, Egger C, Held U, Jackisch C. The Effect of Collaborative Reviews of Electronic Patient-Reported Outcomes on the Congruence of Patient- and Clinician-Reported Toxicity in Cancer Patients Receiving Systemic Therapy: Prospective, Multicenter, Observational Clinical Trial. J Med Internet Res. 2021 Aug 5;23(8):e29271. doi: 10.2196/29271. PMID 34383675
- [Derived] Trojan A, Battig B, Mannhart M, Seifert B, Brauchbar MN, Egbring M. Effect of Collaborative Review of Electronic Patient-Reported Outcomes for Shared Reporting in Breast Cancer Patients: Descriptive Comparative Study. JMIR Cancer. 2021 Mar 17;7(1):e26950. doi: 10.2196/26950. PMID 33729162